CLINICAL TRIAL: NCT01703208
Title: A Randomized, Double-blind, Placebo-controlled, Multicenter Study to Assess Cardiovascular Outcomes Following Treatment With MK-3102 in Subjects With Type 2 Diabetes Mellitus
Brief Title: A Study to Assess Cardiovascular Outcomes Following Treatment With Omarigliptin (MK-3102) in Participants With Type 2 Diabetes Mellitus (MK-3102-018)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The study was terminated for business reasons and not due to any safety or efficacy concerns related to omarigliptin
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 3102-018; 2012-002414-39 (EudraCT Number); MK-3102-018 (Other: Merck study number)
Record Dates: First submitted 2012-10-05; First posted 2012-10-10 (Estimated); Results first posted 2017-12-12 (Actual); Last update posted 2018-11-06 (Actual); Status verified 2018-10

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — 2-(2,5-difluorophenyl)-5-(2-(methylsulfonyl)-2,6-dihydropyrrolo(3,4-c)pyrazol-5(4H)-yl)tetrahydro-2H-pyran-3-amine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Omarigliptin (Experimental): Omarigliptin (MK-3102) 25 mg capsule or tablet administered orally once weekly
  Interventions: Drug: Omarigliptin
- Placebo (Placebo Comparator): Matching placebo to omarigliptin capsule or tablet administered orally once weekly
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Omarigliptin — Omarigliptin (MK-3102) 25 mg capsule or tablet administered orally once weekly
  Arms: Omarigliptin
Drug: Placebo — Matching placebo to omarigliptin capsule or tablet administered orally once weekly
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the cardiovascular (CV) safety profile of omarigliptin in participants with type 2 diabetes mellitus (T2DM). The primary hypothesis is that treatment with omarigliptin 25 mg once weekly is non-inferior to treatment with placebo and active comparators across the omarigliptin program with regard to the risk of developing a confirmed event in the primary CV composite endpoint.

DETAILED DESCRIPTION:
The trial was amended to extend the length of the trial in order to meet FDA requirements for the post-approval assessment of cardiovascular (CV) safety. The trial now contains 2 time intervals: Period 1 and Period 2. Period 1 refers to the time interval up to this recent protocol amendment and Period 2, the time interval from this protocol amendment until the end of the study. Participants in Period 1 will be re-consented and continue into Period 2. If required, additional participants will be enrolled in Period 2. Stage 1 refers to the prefiling United States Food and Drug Administration (US FDA) requirement to rule out a 80% increased CV risk. Stage 2 refers to the US FDA post-marketing requirement to rule out a 30% increased CV risk. The Stage 1 assessment of CV risk occurred during Period 1 and was based on a meta-analysis of major adverse CV events (MACE) and unstable angina across the omarigliptin Phase 2/Phase 3 program. The Stage 2 assessment will be based on MACE in P018 alone including CV events from both Period 1 and Period 2.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with type 2 diabetes mellitus
* Is on one of the following diabetes treatment regimens that is stable for at least 12 weeks (except for pioglitazone for at least 16 weeks) and is within the associated A1C range for that treatment regimen:

  1. A1C >= 6.5% and <= 10.0% (>=48 mmol/mol and <=86 mmol/mol) on: (a) diet or exercise alone (not on antihyperglycemic agent [AHA] for >= 12 weeks) OR (b) monotherapy with metformin (MF), pioglitazone (PIO) or an alpha-glucosidase inhibitor (AGI) or a sodium-glucose cotransporter inhibitor (SGLT2i) OR (c) dual combination therapy with MF, PIO, AGI or SGLT2i OR
  2. A1C >= 7.0% and <=10.0% (>=53 mmol/mol and <=86 mmol/mol) on (a) monotherapy with a sulfonylurea or meglitinide OR (b) dual combination therapy with a sulfonylurea or a meglitinide and MF, PIO, AGI, or SGLT2i OR
  3. A1C >=7.0% and <=10.0% (>=53 mmol/mol and <=86 mmol/mol) on one of the following insulin regimens (with or without metformin): (a) basal insulin (e.g.; insulin glargine, insulin detemir, NPH insulin, degludec) OR (b) prandial insulin (e.g. regular, aspart, lispro, glulisine) OR (c) basal/prandial insulin regimen consisting of multiple dose insulin injections of basal and prandial insulin or the use of pre-mixed insulin (e.g., Novolog 70/30®, Novolin 70/30®, Humalog 75/25®, or Humulin 70/30®
* Pre-existing vascular disease (coronary artery disease, ischemic cerebrovascular disease, atherosclerotic peripheral artery disease)
* (1) Male; (2) female not of reproductive potential; or (3) female of reproductive potential who agrees to remain abstinent or use alone or in conjunction with their partner 2 methods of contraception to prevent pregnancy during the study and for 21 days after the last dose of study drug.

Exclusion Criteria:

* History of type 1 diabetes mellitus or a history of ketoacidosis
* Treated with rosiglitazone, a dipeptidyl peptidase-IV (DPP-4) inhibitor, or a glucagon-like peptide-1 (GLP-1) receptor agonist within 12 weeks prior to study participation or previously treated with omarigliptin
* On a weight loss program and is not in the maintenance phase or has been on a weight loss medication in the past 6 months or has undergone bariatric surgery within 12 months prior to study participation
* Medical history of active liver disease (other than non-alcoholic hepatic steatosis), including chronic active hepatitis B or C, primary biliary cirrhosis, or symptomatic gallbladder disease
* Human immunodeficiency virus (HIV) as assessed by medical history
* New or worsening coronary heart disease, congestive heart failure, myocardial infarction, unstable angina, coronary artery intervention, stroke, or transient ischemic neurological disorder within the past 3 months
* History of malignancy <=5 years prior to study participation, except for adequately treated basal cell or squamous cell skin cancer, or in situ cervical cancer
* Clinically important hematological disorder (such as aplastic anemia, myeloproliferative or myelodysplastic syndromes, thrombocytopenia)
* Pregnant or breast feeding, or is expecting to conceive or donate eggs during the trial, including 21 days following the last dose of study drug

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4202 (Actual)
Dates: Start 2012-10-05 (Actual); Primary Completion 2016-05-13 (Actual); Study Completion 2017-03-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Gantz I, Chen M, Suryawanshi S, Ntabadde C, Shah S, O'Neill EA, Engel SS, Kaufman KD, Lai E. A randomized, placebo-controlled study of the cardiovascular safety of the once-weekly DPP-4 inhibitor omarigliptin in patients with type 2 diabetes mellitus. Cardiovasc Diabetol. 2017 Sep 11;16(1):112. doi: 10.1186/s12933-017-0593-8. PMID 28893244

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 559 sites received IEC/IRB approval in 40 countries and 547 were shipped clinical supplies. Of the 559 sites, 525 screened at least 1 participant.
  An insulin sub-study of MK-3102-018 was performed and included the sub-population of participants receiving ≥20 units/day of background insulin with or without metformin.
Pre-assignment Details: On April 8, 2016, Merck & Co. Inc. announced that it would not submit marketing applications for omarigliptin (MK-3102) in the US and Europe for business reasons only. Because of this decision, the MK-3102-018 study was terminated early on May 13, 2016. Due to delays in study close-out the Last-Participant-Last-Visit occurred on March 22, 2017.
Groups:
- Omarigliptin 25 mg: Omarigliptin (MK-3102) 25 mg capsule or tablet administered orally once weekly
- Placebo: Matching placebo to omarigliptin capsule or tablet administered once weekly.
Period: Overall Study
Arm/Group | Omarigliptin 25 mg | Placebo
Started | 2100 | 2102
Treated | 2092 | 2100
Completed | 0 | 0
Not Completed | 2100 | 2102
Not completed — Death | 61 | 48
Not completed — Lack of Efficacy | 1 | 2
Not completed — Lost to Follow-up | 68 | 62
Not completed — Non-Compliance with Study Drug | 1 | 0
Not completed — Excluded Medication | 1 | 2
Not completed — Site Discontinued Study Participation | 23 | 27
Not completed — Physician Decision | 11 | 13
Not completed — Progressive disease | 2 | 2
Not completed — Protocol Violation | 1 | 1
Not completed — Study Terminated by Sponsor | 1710 | 1716
Not completed — Withdrawal by Subject | 205 | 209
Not completed — Adverse Event | 14 | 19
Not completed — Technical Problems | 0 | 1
Not completed — Protocol Deviation | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Omarigliptin 25 mg | Placebo | Total
Number analyzed (Participants) | 2100 | 2102 | 4202
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.7 (8.5) | 63.6 (8.5) | 63.6 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 639 | 615 | 1254
  Male | 1461 | 1487 | 2948
Hemoglobin A1C % [Mean (Standard Deviation); unit: Percent] — Hemoglobin A1C is blood marker used to report average blood glucose levels over prolonged periods of time and is reported as a percentage (%).
  Percent | 7.99 (0.86) | 8.03 (0.89) | 8.01 (0.87)
Fasting Plasma Glucose (FPG) [Mean (Standard Deviation); unit: mg/dL] | 184.1 (52.2) | 179.5 (45.7) | 180.4 (47.8)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With MACE-plus (Confirmed Cardiovascular [CV]-Related Death, Nonfatal Myocardial Infarction [MI], Nonfatal Stroke, or Hospitalization Due to Unstable Angina)
Description: Participants with confirmed MACE-plus events (confirmed cardiovascular, CV-related death, nonfatal myocardial infarction [MI], nonfatal stroke, or hospitalization due to unstable angina). In the MK-3102-018 study, MACE plus events had a data cut-off date of April 15, 2015.
Time Frame: Up to 156 weeks
Population: The analysis population included all randomized participants who took at least one dose of blinded study medication and were evaluated for MACE-plus events.
Measure: Number; unit: Participants
Arm/Group | Omarigliptin 25 mg | Placebo
Number analyzed (Participants) | 2090 | 2100
Participants | 66 [-1.14 to -0.90] | 70 [-1.20 to -0.96]

2. Primary Outcome: Number of Participants With an Event of MACE (Confirmed CV-Related Death, Fatal and Nonfatal MI, and Fatal and Nonfatal Stroke)
Description: Participants with an Event of MACE (confirmed cardiovascular, CV-related death, fatal and nonfatal myocardial infarction [MI], and fatal and nonfatal stroke).
Time Frame: Up to 179 weeks
Population: The analysis population included all randomized participants who took at least one dose of blinded trial medication.
Measure: Number; unit: Participants
Arm/Group | Omarigliptin 25 mg | Placebo
Number analyzed (Participants) | 2092 | 2100
Participants | 114 [-1.14 to -0.90] | 114 [-1.20 to -0.96]

3. Primary Outcome: Number of Participants With an Event Per 100 Person-Years for First Event of MACE (Confirmed CV-Related Death, Fatal and Nonfatal MI, and Fatal and Nonfatal Stroke)
Description: Participants with an event of MACE (confirmed cardiovascular, CV-related death, fatal and nonfatal myocardial infarction [MI], and fatal and nonfatal stroke). Person-years were calculated as the sum of all participants' follow-up time to first event.
Time Frame: Up to 179 weeks
Population: The analysis population included all randomized participants who took at least one dose of blinded trial medication.
Measure: Number; unit: Participants/100 Person-years
Arm/Group | Omarigliptin 25 mg | Placebo
Number analyzed (Participants) | 2092 | 2100
Participants/100 Person-years | 2.96 [-1.14 to -0.90] | 2.97 [-1.20 to -0.96]
Statistical Analysis 1: Comparison: Omarigliptin 25 mg vs Placebo; Test type: Superiority or Other; Hazard Ratio (HR) = 1.00, 95% CI 2-sided [0.77 to 1.29] — Based on the proportional hazards model that includes treatment as an explanatory factor

4. Primary Outcome: Change From Baseline in Hemoglobin A1C (A1C) at Week 18
Description: A1C is blood marker used to report average blood glucose levels over prolonged periods of time and is reported as a percentage (%). This change from baseline reflects the Week 18 A1C minus the Week 0 A1C.
Time Frame: Baseline and Week 18
Population: The analysis population consisted of all randomized participants who received at least one dose of blinded study medication and had a baseline or a post-randomization measurement.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent
Arm/Group | Omarigliptin 25 mg | Placebo
Number analyzed (Participants) | 2092 | 2100
Percent | -0.58 (0.82) [-0.62 to -0.55] | -0.16 (0.88) [-0.19 to -0.12]
Statistical Analysis 1: Comparison: Omarigliptin 25 mg vs Placebo; Test type: Superiority or Other; Difference in the least squares means = -0.43, 95% CI 2-sided [-0.48 to -0.37]

5. Primary Outcome: Change From Baseline in A1C at Week 18 in a Sub-Study of Participants Taking Insulin (With or Without Metformin)
Description: as for outcome 4
Time Frame: Baseline and Week 18
Population: The analysis population consists of all randomized participants in a sub-study of participants taking insulin who received at least one dose of blinded study medication and had a baseline or a post-randomization measurement.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage
Arm/Group | Omarigliptin 25 mg | Placebo
Number analyzed (Participants) | 535 | 509
Percentage | -0.50 [-0.57 to -0.42] | -0.11 [-0.19 to -0.03]
Statistical Analysis 1: Comparison: Omarigliptin 25 mg vs Placebo; Test type: Superiority or Other; p < 0.001, Longitudinal data analysis; Longitudinal data analysis model including terms for treatment, time and the interaction of time by treatment; Difference in the LS Means vs Placebo = -0.39, 95% CI 2-sided [-0.50 to -0.27]

6. Primary Outcome: Percentage of Participants Who Experienced at Least One Adverse Event in a Sub-study of Participants Taking Insulin Excluding Data After Background Antihyperglycemic Agent (AHA) Change
Description: An AE is defined as any unfavorable and unintended sign including an abnormal laboratory finding, symptom or disease associated with the use of a medical treatment or procedure, regardless of whether it is considered related to the medical treatment or procedure, that occurs during the course of the study.
Time Frame: Up to Week 18
Population: The analysis population included all randomized participants in a sub-study of participants taking insulin who received at least one dose of blinded study medication.
Measure: Number; unit: Percentage of participants
Arm/Group | Omarigliptin 25 mg | Placebo
Number analyzed (Participants) | 535 | 509
Percentage of participants | 48.8 | 49.9
Statistical Analysis 1: Comparison: Omarigliptin 25 mg vs Placebo; Test type: Superiority or Other; Difference in Percent vs. Placebo = -1.1, 95% CI 2-sided [-7.2 to 4.9] — Based on Miettinen & Nurminen method. The 95% CI was computed only for those endpoints with at least 4 participants having events in one or more treatment groups

7. Primary Outcome: Percentage of Participants Who Discontinued From Study Drug Due to an Adverse Event in a Sub-Study of Participants Taking Insulin Excluding Data After Background AHA Change
Description: as for outcome 6
Time Frame: Up to Week 18
Population: as for outcome 6
Measure: Number; unit: Percentage of participants
Arm/Group | Omarigliptin 25 mg | Placebo
Number analyzed (Participants) | 535 | 509
Percentage of participants | 1.1 [-3.13 to -2.25] | 0.8 [-4.18 to -3.29]
Statistical Analysis 1: Comparison: Omarigliptin 25 mg vs Placebo; Test type: Superiority or Other; Difference in Percentage vs. Placebo = 0.3, 95% CI 2-sided [-1.0 to 1.7] — [estimate comment as in outcome 6, analysis 1]

8. Secondary Outcome: Number of Participants With an Event of CV-Related Death
Description: Participants with adjudicated and confirmed AEs of cardiovascular-related death.
Time Frame: Up to 179 weeks
Population: The analysis population consisted of all randomized participants who received at least one dose of blinded study medication.
Measure: Number; unit: Participants
Arm/Group | Omarigliptin 25 mg | Placebo
Number analyzed (Participants) | 2092 | 2100
Participants | 37 [-40.04 to -31.42] | 35 [-41.21 to -32.62]

9. Secondary Outcome: Number of Participants With an Event Per 100 Person-Years of CV-Related Death
Description: Participants with adjudicated and confirmed AEs of cardiovascular-related death. Person-years were calculated as the sum of all participants' follow-up time to event.
Time Frame: Up to 179 weeks
Population: The analysis population consisted of all participants who took at least one dose of blinded study medication.
Measure: Number; unit: Participants/100 person-years
Arm/Group | Omarigliptin 25 mg | Placebo
Number analyzed (Participants) | 2092 | 2100
Participants/100 person-years | 0.94 [-40.04 to -31.42] | 0.89 [-41.21 to -32.62]
Statistical Analysis 1: Comparison: Omarigliptin 25 mg vs Placebo; Test type: Superiority or Other; Hazard Ratio (HR) = 1.06, 95% CI 2-sided [0.66 to 1.68] — Based on the proportional hazards model that includes treatment as an explanatory factor

10. Secondary Outcome: Number of Participants With an Event of First MI (Fatal and Non-fatal)
Description: Participants with adjudicated and confirmed AEs of fatal and non-fatal MI.
Time Frame: Up to 179 weeks
Population: The analysis population consisted of all participants who took at least one dose of blinded study medication.
Measure: Number; unit: Participants
Arm/Group | Omarigliptin 25 mg | Placebo
Number analyzed (Participants) | 2092 | 2100
Participants | 52 [-40.04 to -31.42] | 60 [-41.21 to -32.62]

11. Secondary Outcome: Number of Participants With an Event Per 100 Person-Years of First MI (Fatal and Non-fatal)
Description: Participants with adjudicated and confirmed AEs of fatal and non-fatal MI. Person-years were calculated as the sum of all participants' follow-up time to first event.
Time Frame: Up to 179 weeks
Population: The analysis population consisted of all participants who took at least one dose of blinded study medication.
Measure: Number; unit: Participants/100 person-years
Arm/Group | Omarigliptin 25 mg | Placebo
Number analyzed (Participants) | 2092 | 2100
Participants/100 person-years | 1.34 [-40.04 to -31.42] | 1.55 [-41.21 to -32.62]
Statistical Analysis 1: Comparison: Omarigliptin 25 mg vs Placebo; Test type: Superiority or Other; Hazard Ratio (HR) = 0.87, 95% CI 2-sided [0.60 to 1.26] — Based on the proportional hazards model that includes treatment as an explanatory factor

12. Secondary Outcome: Number of Participants With an Event of Stroke (Fatal and Non-fatal)
Description: Participants with adjudicated and confirmed AEs fatal and non-fatal stroke.
Time Frame: Up to 179 weeks
Population: The analysis population consisted of all participants who took at least one dose of blinded study medication.
Measure: Number; unit: Participants
Arm/Group | Omarigliptin 25 mg | Placebo
Number analyzed (Participants) | 2092 | 2100
Participants | 32 [-40.04 to -31.42] | 34 [-41.21 to -32.62]

13. Secondary Outcome: Number of Participants With an Event Per 100 Person-Years of First Stroke (Fatal and Non-fatal)
Description: Participants with adjudicated and confirmed AEs fatal and non-fatal stroke. Person-years were calculated as the sum of all participants' follow-up time to event.
Time Frame: Up to 179 weeks
Population: The analysis population consisted of all participants who took at least one dose of blinded study medication.
Measure: Number; unit: Participants/100 person-years
Arm/Group | Omarigliptin 25 mg | Placebo
Number analyzed (Participants) | 2092 | 2100
Participants/100 person-years | 0.82 [-40.04 to -31.42] | 0.88 [-41.21 to -32.62]
Statistical Analysis 1: Comparison: Omarigliptin 25 mg vs Placebo; Test type: Superiority or Other; Hazard Ratio (HR) = 0.94, 95% CI 2-sided [0.58 to 1.52] — Based on the proportional hazards model that includes treatment as an explanatory factor

14. Secondary Outcome: Number of Participants With an Event of All-Cause Death
Description: All-cause death was death from any cause.
Time Frame: Up to 179 weeks
Population: The analysis population included all randomized participants who took at least one dose of blinded trial medication.
Measure: Number; unit: Participants
Arm/Group | Omarigliptin 25 mg | Placebo
Number analyzed (Participants) | 2092 | 2100
Participants | 64 | 50

15. Secondary Outcome: Number of Participants With an Event Per 100 Person-Years of the Event of All-Cause Death
Description: All-cause death was death for any cause. Person-years were calculated as the sum of all participants' follow-up time to event.
Time Frame: Up to 179 weeks
Population: The analysis population included all randomized participants who took at least one dose of blinded study medication.
Measure: Number; unit: Participants/100 Person-years
Arm/Group | Omarigliptin 25 mg | Placebo
Number analyzed (Participants) | 2092 | 2100
Participants/100 Person-years | 1.63 | 1.28
Statistical Analysis 1: Comparison: Omarigliptin 25 mg vs Placebo; Test type: Superiority or Other; Hazard Ratio (HR) = 1.28, 95% CI 2-sided [0.88 to 1.85] — Based on the proportional hazards model that includes treatment as an explanatory factor

16. Secondary Outcome: Change From Baseline in A1C at Week 142
Description: A1C is blood marker used to report average blood glucose levels over prolonged periods of time and is reported as a percentage (%). This change from baseline reflects the Week 142 A1C minus the Week 0 A1C.
Time Frame: Baseline and Week 142
Population: as for outcome 4
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent
Arm/Group | Omarigliptin 25 mg | Placebo
Number analyzed (Participants) | 2092 | 2100
Percent | -0.36 (0.06) [-0.47 to -0.25] | -0.06 (1.12) [-0.17 to 0.05]
Statistical Analysis 1: Comparison: Omarigliptin 25 mg vs Placebo; Test type: Superiority or Other; Difference in the Least Squares Means = -0.30, 95% CI 2-sided [-0.46 to -0.14] — Longitudinal Data Analysis (LDA) model including terms for treatment, time, and the interaction of time by treatment

17. Secondary Outcome: Percentage of Participants Achieving a Target A1C <7.0 % (53 mmol/Mol) at 4 Months
Description: A1C is blood marker used to report average blood glucose levels over prolonged periods of time and is reported as a percentage (%).
Time Frame: 4 months
Population: Data for this efficacy endpoint was not collected, analyzed or summarized.
Arm/Group | Omarigliptin 25 mg | Placebo
Number analyzed (Participants) | 0 | 0

18. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG) at 4 Months
Description: This change from baseline reflects the Month 4 FPG minus the Week 0 FPG.
Time Frame: Baseline and 4 months
Population: Data for this efficacy endpoint was not collected, analyzed or summarized.
Arm/Group | Omarigliptin 25 mg | Placebo
Number analyzed (Participants) | 0 | 0

19. Secondary Outcome: Time to Initiation of Long-Term Insulin Therapy in Participants Not Receiving Insulin at Baseline
Description: Long-term insulin therapy was defined as a continuous period of insulin use of more than 3 months.
Time Frame: Up to 179 weeks
Population: Data for this efficacy endpoint was not collected, analyzed or summarized.
Arm/Group | Omarigliptin 25 mg | Placebo
Number analyzed (Participants) | 0 | 0

20. Secondary Outcome: Percentage of Participants Who Experienced at Least One Adverse Event
Description: as for outcome 6
Time Frame: Up to 234 weeks
Population: The analysis population included all randomized participants who took at least one dose of blinded study medication.
Measure: Number; unit: Percentage of participants
Arm/Group | Omarigliptin 25 mg | Placebo
Number analyzed (Participants) | 2092 | 2100
Percentage of participants | 78.3 | 76.8

21. Secondary Outcome: Percentage of Participants Who Discontinued From Study Drug Due to an Adverse Event
Description: as for outcome 6
Time Frame: Up to 212 weeks
Population: The analysis population included all randomized participants who took at least one dose of blinded study medication.
Measure: Number; unit: Percentage of participants
Arm/Group | Omarigliptin 25 mg | Placebo
Number analyzed (Participants) | 2092 | 2100
Percentage of participants | 4.1 | 3.6

22. Secondary Outcome: Change From Baseline in FPG at Week 18 in a Sub-Study of Participants Taking Insulin
Description: This change from baseline reflects the Week 18 FPG minus the Week 0 FPG.
Time Frame: Baseline and Week 18
Population: The analysis population consisted of all randomized participants in a sub-study of participants taking insulin who received at least one dose of blinded study medication and had a baseline or a post-randomization measurement.
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Omarigliptin 25 mg | Placebo
Number analyzed (Participants) | 535 | 509
mg/dL | -6.8 [-12.1 to -1.5] | -3.6 [-9.1 to 1.8]
Statistical Analysis 1: Comparison: Omarigliptin 25 mg vs Placebo; Test type: Superiority or Other; p = 0.421, Longitudinal constrained data analysis; Difference in the least squares means = -3.1, 95% CI 2-sided [-10.8 to 4.5] — Based on a LDA model including terms for treatment, time and the interaction of time by treatment

23. Secondary Outcome: Percentage of Participants Achieving a Target A1C <7.0 % (53 mmol/Mol) at Week 18 in a Sub-Study of Participants Taking Insulin
Description: A1C is blood marker used to report average blood glucose levels over prolonged periods of time and is reported as a percentage (%). Analysis was performed with multiple data imputation.
Time Frame: 18 weeks
Population: The analysis population consisted of all randomized participants in a sub-study of participants taking insulin who received at least one dose of blinded study medication.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Omarigliptin 25 mg | Placebo
Number analyzed (Participants) | 535 | 509
Percentage of participants | 22.0 [18.5 to 26.1] | 10.2 [7.5 to 13.6]
Statistical Analysis 1: Comparison: Omarigliptin 25 mg vs Placebo; Test type: Superiority or Other; p < 0.001, Miettinen & Nurminen method — Estimated using standard multiple imputation techniques; Between group rate difference = 11.9, 95% CI 2-sided [6.9 to 16.8]

24. Other Pre Specified Outcome: Number of Participants With an Event of First Hospitalization for Heart Failure (Exploratory)
Description: Participants with adjudicated and confirmed events of first hospitalization for heart failure.
Time Frame: Up to 179 weeks
Population: The analysis population consisted of all participants who took at least one dose of blinded study medication.
Measure: Number; unit: Participants
Arm/Group | Omarigliptin 25 mg | Placebo
Number analyzed (Participants) | 2092 | 2100
Participants | 20 | 33

25. Other Pre Specified Outcome: Number of Participants With an Event Per 100 Person-years of the Event of the First Hospitalization for Heart Failure (Exploratory)
Description: Participants with adjudicated and confirmed events of first hospitalization for heart failure. Person-years were calculated as the sum of all participants' follow-up time to event.
Time Frame: Up to 179 weeks
Population: The analysis population consisted of all participants who took at least one dose of blinded study medication.
Measure: Number; unit: Participants/100 Person-years
Arm/Group | Omarigliptin 25 mg | Placebo
Number analyzed (Participants) | 2092 | 2100
Participants/100 Person-years | 0.51 | 0.85
Statistical Analysis 1: Comparison: Omarigliptin 25 mg vs Placebo; Test type: Superiority or Other; Hazard Ratio (HR) = 0.60, 95% CI 2-sided [0.35 to 1.05] — Based on the proportional hazards model that includes treatment as an explanatory factor

ADVERSE EVENTS:
Time Frame: Up to 234 weeks
Description: Participants with serious adverse events with an incidence > 0% and with >5% non-serous adverse events in one or more treatment groups during the Treatment Period + Post-Treatment Follow-up including Post-21 days after last dose of blinded study treatment for randomized participants receiving one or more doses of study treatment.
Arm/Group | Omarigliptin 25 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 512/2092 | 503/2100
Other Adverse Events (participants affected / at risk) | 788/2092 | 794/2100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Omarigliptin 25 mg (N=2092) | Placebo (N=2100)
Agranulocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 6 (6) | 4 (4)
Coagulation factor deficiency (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 0 (0) | 2 (3)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Lymphadenitis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Splenic infarction (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Thrombocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 3 (3) | 7 (7)
Acute myocardial infarction (Cardiac disorders) | 30 (35) | 27 (28)
Angina pectoris (Cardiac disorders) | 27 (29) | 31 (36)
Angina unstable (Cardiac disorders) | 33 (39) | 42 (46)
Aortic valve stenosis (Cardiac disorders) | 5 (5) | 1 (1)
Arteriosclerosis coronary artery (Cardiac disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 14 (14) | 16 (17)
Atrial flutter (Cardiac disorders) | 5 (7) | 3 (3)
Atrial tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Atrioventricular block (Cardiac disorders) | 1 (1) | 1 (1)
Atrioventricular block complete (Cardiac disorders) | 3 (3) | 0 (0)
Bradyarrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 2 (2) | 1 (1)
Cardiac aneurysm (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 9 (9) | 4 (4)
Cardiac failure (Cardiac disorders) | 17 (21) | 12 (12)
Cardiac failure acute (Cardiac disorders) | 6 (6) | 4 (4)
Cardiac failure chronic (Cardiac disorders) | 7 (8) | 3 (3)
Cardiac failure congestive (Cardiac disorders) | 14 (16) | 20 (25)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 3 (3)
Cardiogenic shock (Cardiac disorders) | 2 (2) | 4 (4)
Cardiomyopathy (Cardiac disorders) | 0 (0) | 2 (2)
Cardiopulmonary failure (Cardiac disorders) | 1 (1) | 4 (5)
Conduction disorder (Cardiac disorders) | 1 (1) | 0 (0)
Cor pulmonale (Cardiac disorders) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 22 (24) | 23 (24)
Coronary artery insufficiency (Cardiac disorders) | 0 (0) | 1 (1)
Coronary artery occlusion (Cardiac disorders) | 3 (3) | 4 (4)
Coronary artery stenosis (Cardiac disorders) | 9 (9) | 6 (6)
Ischaemic cardiomyopathy (Cardiac disorders) | 1 (1) | 1 (1)
Left ventricular failure (Cardiac disorders) | 1 (1) | 2 (2)
Myocardial infarction (Cardiac disorders) | 19 (19) | 17 (19)
Myocardial ischaemia (Cardiac disorders) | 5 (6) | 3 (3)
Myocardial reperfusion injury (Cardiac disorders) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1)
Right ventricular failure (Cardiac disorders) | 1 (1) | 0 (0)
Silent myocardial infarction (Cardiac disorders) | 2 (2) | 1 (1)
Sinus node dysfunction (Cardiac disorders) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 3 (4) | 1 (1)
Ventricular arrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular extrasystoles (Cardiac disorders) | 1 (1) | 3 (3)
Ventricular fibrillation (Cardiac disorders) | 3 (3) | 0 (0)
Ventricular tachyarrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 2 (2) | 3 (4)
Congenital claw toe (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Encephalocele (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Deafness neurosensory (Ear and labyrinth disorders) | 0 (0) | 2 (2)
Deafness unilateral (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 2 (2) | 0 (0)
Vertigo positional (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Vestibular disorder (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Goitre (Endocrine disorders) | 1 (1) | 1 (1)
Cataract (Eye disorders) | 0 (0) | 2 (2)
Keratitis (Eye disorders) | 1 (1) | 0 (0)
Retinal detachment (Eye disorders) | 0 (0) | 2 (3)
Retinal haemorrhage (Eye disorders) | 0 (0) | 1 (1)
Retinal tear (Eye disorders) | 1 (1) | 0 (0)
Vitreous haemorrhage (Eye disorders) | 0 (0) | 2 (2)
Abdominal hernia (Gastrointestinal disorders) | 2 (2) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Acquired oesophageal web (Gastrointestinal disorders) | 1 (1) | 0 (0)
Anal spasm (Gastrointestinal disorders) | 0 (0) | 1 (1)
Chronic gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Crohn's disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diabetic gastroenteropathy (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diabetic gastroparesis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Diverticular perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diverticulum (Gastrointestinal disorders) | 0 (0) | 1 (1)
Duodenal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Enterovesical fistula (Gastrointestinal disorders) | 1 (1) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastric polyps (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 2 (2) | 1 (1)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 2 (2) | 1 (1)
Gastric varices haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastritis erosive (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastroduodenitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 (2) | 2 (2)
Gastrointestinal ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ileus paralytic (Gastrointestinal disorders) | 1 (1) | 1 (1)
Impaired gastric emptying (Gastrointestinal disorders) | 1 (1) | 0 (0)
Incarcerated umbilical hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 5 (6) | 2 (2)
Intestinal obstruction (Gastrointestinal disorders) | 2 (2) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 1 (1) | 4 (4)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 2 (3)
Noninfective gingivitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 3 (3) | 0 (0)
Pancreatic cyst (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 2 (2) | 1 (1)
Pancreatitis chronic (Gastrointestinal disorders) | 0 (0) | 1 (1)
Peptic ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 2 (2)
Retroperitoneal haematoma (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 2 (2)
Strangulated umbilical hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 3 (3)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Cardiac death (General disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 6 (8) | 1 (1)
Complication associated with device (General disorders) | 2 (2) | 1 (1)
Death (General disorders) | 4 (4) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 5 (5) | 1 (1)
Non-cardiac chest pain (General disorders) | 5 (5) | 8 (10)
Sudden cardiac death (General disorders) | 0 (0) | 4 (4)
Sudden death (General disorders) | 6 (6) | 3 (3)
Vascular stent restenosis (General disorders) | 2 (2) | 1 (1)
Bile duct stone (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholangitis (Hepatobiliary disorders) | 1 (1) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 7 (7) | 3 (3)
Cholecystitis acute (Hepatobiliary disorders) | 4 (4) | 4 (4)
Cholecystitis chronic (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 5 (5) | 3 (3)
Hepatic cirrhosis (Hepatobiliary disorders) | 0 (0) | 2 (2)
Hepatorenal syndrome (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hydrocholecystis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Jaundice (Hepatobiliary disorders) | 1 (1) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 1 (1) | 1 (1)
Abdominal abscess (Infections and infestations) | 2 (2) | 0 (0)
Abscess intestinal (Infections and infestations) | 1 (1) | 0 (0)
Abscess limb (Infections and infestations) | 2 (2) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 2 (2)
Atypical pneumonia (Infections and infestations) | 1 (1) | 1 (1)
Bacterial sepsis (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 6 (6) | 2 (2)
Bronchitis viral (Infections and infestations) | 0 (0) | 1 (1)
Bronchopulmonary aspergillosis (Infections and infestations) | 1 (1) | 0 (0)
Bronchopulmonary aspergillosis allergic (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 11 (11) | 2 (3)
Chronic hepatitis C (Infections and infestations) | 1 (1) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 1 (1)
Diabetic foot infection (Infections and infestations) | 0 (0) | 1 (1)
Diabetic gangrene (Infections and infestations) | 1 (1) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (1) | 1 (1)
Endocarditis bacterial (Infections and infestations) | 0 (0) | 1 (1)
Endophthalmitis (Infections and infestations) | 1 (1) | 0 (0)
Enterococcal sepsis (Infections and infestations) | 1 (1) | 0 (0)
Epididymitis (Infections and infestations) | 1 (1) | 0 (0)
Erysipelas (Infections and infestations) | 1 (1) | 2 (2)
Escherichia urinary tract infection (Infections and infestations) | 0 (0) | 3 (3)
Febrile infection (Infections and infestations) | 1 (1) | 0 (0)
Fungal infection (Infections and infestations) | 0 (0) | 1 (1)
Gangrene (Infections and infestations) | 6 (7) | 4 (4)
Gas gangrene (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 3 (4) | 3 (3)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 1 (1)
HIV infection (Infections and infestations) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 1 (1)
Infectious pleural effusion (Infections and infestations) | 2 (2) | 0 (0)
Infective exacerbation of bronchiectasis (Infections and infestations) | 1 (1) | 0 (0)
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 1 (1) | 0 (0)
Kidney infection (Infections and infestations) | 0 (0) | 1 (1)
Klebsiella sepsis (Infections and infestations) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 2 (2)
Lung infection (Infections and infestations) | 1 (1) | 0 (0)
Mediastinitis (Infections and infestations) | 1 (1) | 0 (0)
Neuroborreliosis (Infections and infestations) | 1 (1) | 0 (0)
Nosocomial infection (Infections and infestations) | 1 (1) | 0 (0)
Osteomyelitis (Infections and infestations) | 2 (2) | 1 (1)
Paronychia (Infections and infestations) | 0 (0) | 2 (2)
Parotitis (Infections and infestations) | 0 (0) | 1 (1)
Pelvic sepsis (Infections and infestations) | 1 (1) | 0 (0)
Perirectal abscess (Infections and infestations) | 1 (1) | 0 (0)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 35 (37) | 31 (31)
Pneumonia respiratory syncytial viral (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia streptococcal (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia viral (Infections and infestations) | 0 (0) | 1 (1)
Postoperative abscess (Infections and infestations) | 0 (0) | 1 (1)
Pulmonary tuberculosis (Infections and infestations) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 1 (1) | 3 (3)
Pyelonephritis acute (Infections and infestations) | 1 (1) | 1 (1)
Respiratory tract infection (Infections and infestations) | 2 (2) | 0 (0)
Respiratory tract infection viral (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 7 (7) | 5 (5)
Septic shock (Infections and infestations) | 3 (3) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Subdural empyema (Infections and infestations) | 1 (1) | 0 (0)
Tuberculosis (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 2 (2)
Urinary tract infection (Infections and infestations) | 4 (4) | 6 (6)
Urinary tract infection bacterial (Infections and infestations) | 1 (1) | 0 (0)
Urosepsis (Infections and infestations) | 0 (0) | 1 (1)
Viral infection (Infections and infestations) | 2 (2) | 1 (1)
Vulval abscess (Infections and infestations) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 0 (0) | 1 (1)
Acetabulum fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alcohol poisoning (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 3 (3)
Avulsion fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Cardiac procedure complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Chemical peritonitis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 2 (2) | 2 (3)
Coronary artery restenosis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Cystitis radiation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Face injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Fibula fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Flail chest (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Forearm fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Gastrointestinal anastomotic leak (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Incarcerated incisional hernia (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Incisional hernia (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Jaw fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Lower limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Meniscus injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Multiple injuries (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post procedural complication (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Postoperative ileus (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 3 (3)
Road traffic accident (Injury, poisoning and procedural complications) | 3 (3) | 1 (1)
Soft tissue injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Spinal cord injury cervical (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Stomal hernia (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Synovial rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Traumatic haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Vascular graft occlusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0)
Blood glucose increased (Investigations) | 1 (1) | 6 (6)
Blood sodium decreased (Investigations) | 0 (0) | 1 (1)
Heart rate increased (Investigations) | 1 (1) | 0 (0)
Troponin increased (Investigations) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 3 (3)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 3 (3) | 1 (1)
Diabetic metabolic decompensation (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Fluid overload (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Gout (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 5 (5) | 7 (7)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 3 (4) | 5 (5)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Obesity (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Amyotrophy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 2 (2) | 4 (4)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Osteitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 14 (15) | 9 (9)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Periarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 4 (4) | 0 (0)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Trigger finger (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (6) | 10 (15)
Benign neoplasm of eyelid (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Benign renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 5 (5)
Bladder cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Bone cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Breast cancer in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 1 (1)
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Gastrooesophageal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Hepatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 3 (3)
Lung carcinoma cell type unspecified stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 1 (1)
Lung squamous cell carcinoma stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 1 (1)
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastatic gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Neuroendocrine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 1 (1)
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Parathyroid tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 (7) | 4 (4)
Prostate cancer stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Prostate cancer stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Prostatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 3 (3)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 2 (2)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (2)
Small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (3) | 5 (9)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Tonsil cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Urinary tract neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Vocal cord neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Altered state of consciousness (Nervous system disorders) | 0 (0) | 2 (2)
Ataxia (Nervous system disorders) | 1 (1) | 1 (1)
Basal ganglia infarction (Nervous system disorders) | 1 (1) | 0 (0)
Basal ganglia stroke (Nervous system disorders) | 0 (0) | 1 (1)
Brain stem infarction (Nervous system disorders) | 2 (2) | 0 (0)
Carotid artery stenosis (Nervous system disorders) | 4 (4) | 7 (7)
Cauda equina syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 1 (1) | 2 (2)
Cerebral infarction (Nervous system disorders) | 4 (4) | 2 (2)
Cerebral ischaemia (Nervous system disorders) | 0 (0) | 2 (2)
Cerebral small vessel ischaemic disease (Nervous system disorders) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 9 (10) | 9 (9)
Cerebrovascular insufficiency (Nervous system disorders) | 2 (2) | 0 (0)
Cervical radiculopathy (Nervous system disorders) | 0 (0) | 1 (1)
Cervicobrachial syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Coma (Nervous system disorders) | 0 (0) | 1 (1)
Dementia (Nervous system disorders) | 0 (0) | 1 (1)
Dementia Alzheimer's type (Nervous system disorders) | 0 (0) | 1 (1)
Diabetic neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 2 (2)
Embolic stroke (Nervous system disorders) | 1 (1) | 1 (1)
Encephalopathy (Nervous system disorders) | 0 (0) | 2 (2)
Epilepsy (Nervous system disorders) | 1 (1) | 0 (0)
Facial paralysis (Nervous system disorders) | 1 (1) | 0 (0)
Haemorrhagic stroke (Nervous system disorders) | 1 (1) | 2 (2)
Headache (Nervous system disorders) | 1 (1) | 1 (1)
Hypertensive encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
IIIrd nerve paralysis (Nervous system disorders) | 1 (1) | 0 (0)
Intracranial aneurysm (Nervous system disorders) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 11 (11) | 17 (17)
Lacunar infarction (Nervous system disorders) | 2 (2) | 0 (0)
Loss of consciousness (Nervous system disorders) | 1 (1) | 1 (1)
Lumbar radiculopathy (Nervous system disorders) | 0 (0) | 1 (1)
Meralgia paraesthetica (Nervous system disorders) | 1 (1) | 0 (0)
Migraine (Nervous system disorders) | 1 (1) | 0 (0)
Monoparesis (Nervous system disorders) | 0 (0) | 1 (1)
Myelitis transverse (Nervous system disorders) | 0 (0) | 1 (1)
Nerve root compression (Nervous system disorders) | 1 (1) | 0 (0)
Parkinson's disease (Nervous system disorders) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 2 (2)
Radiculopathy (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 7 (8) | 2 (4)
Thalamic infarction (Nervous system disorders) | 1 (1) | 0 (0)
Toxic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 11 (11) | 11 (11)
VIth nerve paralysis (Nervous system disorders) | 0 (0) | 2 (2)
Vascular dementia (Nervous system disorders) | 0 (0) | 1 (1)
Vertebrobasilar insufficiency (Nervous system disorders) | 0 (0) | 2 (2)
Device breakage (Product Issues) | 0 (0) | 1 (1)
Device malfunction (Product Issues) | 0 (0) | 1 (1)
Abnormal behaviour (Psychiatric disorders) | 0 (0) | 1 (1)
Acute stress disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Alcoholism (Psychiatric disorders) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 2 (2) | 3 (3)
Major depression (Psychiatric disorders) | 0 (0) | 2 (2)
Mental disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Panic attack (Psychiatric disorders) | 0 (0) | 1 (1)
Schizophrenia (Psychiatric disorders) | 1 (3) | 0 (0)
Somatic symptom disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Stress (Psychiatric disorders) | 0 (0) | 1 (1)
Substance-induced mood disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Suicide attempt (Psychiatric disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 11 (11) | 6 (6)
Calculus urethral (Renal and urinary disorders) | 1 (1) | 0 (0)
Calculus urinary (Renal and urinary disorders) | 2 (2) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 2 (2) | 0 (0)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Haemorrhage urinary tract (Renal and urinary disorders) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 5 (5) | 2 (2)
Renal colic (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 1 (1)
Stag horn calculus (Renal and urinary disorders) | 1 (1) | 0 (0)
Ureteric stenosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Ureterolithiasis (Renal and urinary disorders) | 2 (2) | 0 (0)
Urethral stenosis (Renal and urinary disorders) | 1 (1) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1) | 1 (1)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 2 (2) | 1 (1)
Breast fibrosis (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Genital prolapse (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Ovarian cyst (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Prostatic dysplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Prostatitis (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Uterine haemorrhage (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Uterine prolapse (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 7 (9) | 5 (6)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 5 (5)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (3)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dermatosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Diabetic foot (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (4)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 6 (6) | 0 (0)
Aortic aneurysm (Vascular disorders) | 2 (2) | 1 (1)
Aortic stenosis (Vascular disorders) | 1 (1) | 2 (2)
Arterial occlusive disease (Vascular disorders) | 0 (0) | 1 (1)
Circulatory collapse (Vascular disorders) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 2 (2) | 3 (4)
Dry gangrene (Vascular disorders) | 2 (2) | 0 (0)
Extremity necrosis (Vascular disorders) | 2 (2) | 2 (2)
Haematoma (Vascular disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 7 (7) | 8 (8)
Hypertensive crisis (Vascular disorders) | 2 (2) | 3 (3)
Hypertensive emergency (Vascular disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Iliac artery occlusion (Vascular disorders) | 1 (1) | 0 (0)
Intermittent claudication (Vascular disorders) | 1 (1) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 1 (1) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 14 (17) | 10 (11)
Peripheral artery occlusion (Vascular disorders) | 0 (0) | 1 (1)
Peripheral artery stenosis (Vascular disorders) | 3 (3) | 2 (2)
Peripheral artery thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Peripheral ischaemia (Vascular disorders) | 1 (2) | 4 (4)
Peripheral vascular disorder (Vascular disorders) | 4 (4) | 1 (1)
Trifascicular block (Cardiac disorders) | 1 (1) | 0 (0)
Catheter site haemorrhage (General disorders) | 0 (0) | 1 (1)
Vascular stent thrombosis (General disorders) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Procedural pneumothorax (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Benign ear neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Ear neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cerebellar infarction (Nervous system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Omarigliptin 25 mg (N=2092) | Placebo (N=2100)
Nasopharyngitis (Infections and infestations) | 123 (167) | 145 (195)
Upper respiratory tract infection (Infections and infestations) | 123 (163) | 120 (150)
Blood glucose increased (Investigations) | 97 (139) | 139 (199)
Hypoglycaemia (Metabolism and nutrition disorders) | 530 (3990) | 473 (3688)
Urinary tract infection (Infections and infestations) | 108 (131) | 98 (141)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the sponsor as confidential must be deleted prior to submission.